CLINICAL TRIAL: NCT05303974
Title: Competency-based Assessment of Ultrasound-guided Joint Injection Skills: A Validity Study
Brief Title: Competency-based Assessment of Ultrasound-guided Joint Injection Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Stine Maya Dreier Carstensen, MD, PhD fellow, Principal investigator, Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2022-003
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Musculoskeletal Diseases
Keywords: Training; Ultrasound; Medical education
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Novices (Experimental): Measurement of competence
  Interventions: Other: Ultrasound guided joint injection
- Intermediates (Experimental): Measurement of competence
  Interventions: Other: Ultrasound guided joint injection
- Experts (Experimental): Measurement of competence
  Interventions: Other: Ultrasound guided joint injection

INTERVENTIONS:
Other: Ultrasound guided joint injection — The participants will perform two ultrasound guided joint injections on a mannequin. The performance of both procedures are videorecorded. All videos will be rated by two blinded raters using the modified IUSE assessment tool.

SUMMARY:
Ultrasound-guided joint injections and aspirations are frequently used in the treatment of rheumatological diseases. Studies have shown that intra-articular glucocorticoid injections (IAGCs) in the early treatment of rheumatoid arthritis is essential and leads to improved disease control and earlier achievement of remission. Unfortunately, many rheumatologists feel insecure performing IAGC due to poor and unstructured training opportunities, which can result in suboptimal treatment and potentially poorer patient outcome.

Nowadays, the gold standard training method has shifted towards competency-based education were objective assessment tools are necessary. A previous study has developed a scale for assessment of invasive ultrasound procedures, the Interventional Ultrasound Skills Evaluation (IUSE) tool. Although expert consensus supports evidence of content validity of the assessment tool, it is not known if the tool can discriminate differences in performance scores between the different levels of experience.

ELIGIBILITY:
Inclusion Criteria:

* Physicians attending the yearly international conference EULAR (Denmark 2022)

  1. Novices: No or little experience with ultrasound guided joint injections.
  2. Intermediates: Participated and completed at least one formal musculoskeletal ultrasound course and performed more than 100 ultrasound guided joint injections.
  3. Experts: Physicians with a long experience with musculoskeletal ultrasound and ultrasound guided joint injections doing the procedure almost daily and providing teaching and/or research within this field.

Exclusion Criteria:

* No informed consent
* Novices/Intermediates: extensive experience with musculoskeletal ultrasound and/or ultrasound guided joint injections.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-29 (Actual); Primary Completion 2022-06-04 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Performance score | Up to 12 months
  Performance score assessed by blinded raters using the modified IUSE assessment tool

CONTACTS AND LOCATIONS:
Overall Officials: Stine Maya D Carstensen, MD, Principal Investigator — Afdeling for Rygkirurgi, Led- og Bindevævssygdomme, COPECARE (Copenhagen Center for Arthritis Research) Rigshospitalet, Glostrup Valdemar Hansens vej 17 2600 Glostrup
Locations (1):
- COPECARE (Copenhagen Center for Arthritis Research), Glostrup Municipality, Denmark

REFERENCES:
- [Result] Kahr Rasmussen N, Nayahangan LJ, Carlsen J, Ekberg O, Brabrand K, Albrecht-Beste E, Nielsen MB, Konge L. Evaluation of competence in ultrasound-guided procedures-a generic assessment tool developed through the Delphi method. Eur Radiol. 2021 Jun;31(6):4203-4211. doi: 10.1007/s00330-020-07280-z. Epub 2020 Nov 17. PMID 33201282
- [Result] Mandl P, Naredo E, Conaghan PG, D'Agostino MA, Wakefield RJ, Bachta A, Backhaus M, Hammer HB, Bruyn GA, Damjanov N, Filippucci E, Grassi W, Iagnocco A, Jousse-Joulin S, Kane D, Koski JM, Moller I, De Miguel E, Schmidt WA, Swen WA, Szkudlarek M, Terslev L, Ziswiler HR, Ostergaard M, Balint PV. Practice of ultrasound-guided arthrocentesis and joint injection, including training and implementation, in Europe: results of a survey of experts and scientific societies. Rheumatology (Oxford). 2012 Jan;51(1):184-90. doi: 10.1093/rheumatology/ker331. Epub 2011 Nov 24. PMID 22120466
- [Result] Hetland ML, Ostergaard M, Ejbjerg B, Jacobsen S, Stengaard-Pedersen K, Junker P, Lottenburger T, Hansen I, Andersen LS, Tarp U, Svendsen A, Pedersen JK, Skjodt H, Ellingsen T, Lindegaard H, Podenphant J, Horslev-Petersen K; CIMESTRA study group. Short- and long-term efficacy of intra-articular injections with betamethasone as part of a treat-to-target strategy in early rheumatoid arthritis: impact of joint area, repeated injections, MRI findings, anti-CCP, IgM-RF and CRP. Ann Rheum Dis. 2012 Jun;71(6):851-6. doi: 10.1136/annrheumdis-2011-200632. Epub 2012 Feb 1. PMID 22302316
- [Result] Bruyn GA, Schmidt WA. How to perform ultrasound-guided injections. Best Pract Res Clin Rheumatol. 2009 Apr;23(2):269-79. doi: 10.1016/j.berh.2008.11.001. PMID 19393570
- [Derived] Carstensen SMD, Just SA, Pfeiffer-Jensen M, Ostergaard M, Konge L, Terslev L. Development and validation of a new tool for assessment of trainees' interventional musculoskeletal ultrasound skills. Rheumatology (Oxford). 2025 Feb 1;64(2):484-492. doi: 10.1093/rheumatology/keae050. PMID 38273715